CLINICAL TRIAL: NCT00644462
Title: Wheeze Detection in Adults During Dynamic Bronchial Situations Measured by PulmoTrack® 2010 With WIM-PC™ Technologies Recording
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: KarmelSonix Ltd. (Industry)
Responsible Party: Dr. Hanna Levy, KarmelSonix Ltd
Other Study IDs: KSI-WZA-01
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Asthma, Bronchial
Keywords: wheeze detection
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Asthmatic subjects
  Interventions: Device: PulmoTrack® 2010 with WIM-PC™ Technologies
- 2: Healthy subjects
  Interventions: Device: PulmoTrack® 2010 with WIM-PC™ Technologies

INTERVENTIONS:
Device: PulmoTrack® 2010 with WIM-PC™ Technologies — wheeze detection during dynamic bronchial situations in infants

SUMMARY:
The PulmoTrack® 2010 with WIM-PC™ Technologies device, indicated for acoustic pulmonary function measurement that quantifies the presence of wheezing. This study was designed in order to evaluate the efficacy and safety of using the WIM-PC™ device for wheeze detection during dynamic bronchial situations in asthmatic adult.

DETAILED DESCRIPTION:
Asthma is defined by the National Asthma Education and Prevention Program (NAEPP) guideline as a 'Chronic inflammatory disorder of the airways in which many cells and cellular elements play a role. The asthma guideline states that inflammation causes recurrent episodes of wheezing, breathlessness and chest tightness that are associated with widespread but variable airflow obstruction.

Wheeze quantification by lung sounds analysis methods is objective, non invasive and has been shown to correlate with clinical status in asthma and bronchiolitis. The recording procedure is simple, requiring only the attachment of 4 ECG-size sensors to the chest wall. A 30-second recording is often adequate to obtain good quality data, where wheezes are detected and counted with high degree of accuracy.

Karmel Sonix Ltd has developed the PulmoTrack® 2010 with WIM-PC™ Technologies device, indicated for acoustic pulmonary function measurement that quantifies the presence of wheezing. This study was designed in order to evaluate the efficacy and safety of using the PulmoTrack® 2010 with WIM-PC™ Technologies device for wheeze detection during dynamic bronchial situations in asthmatic adults.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic or healthy subjects;
* Age 18 and up;
* Not smoking for at the last two years;
* Subject or subject's parents/guardian is able to comprehend and give informed consent for participation in the study.

Exclusion Criteria:

* Chest burns;
* COPD;
* Pregnant or lactating;
* Mechanically ventilatory;
* Homodynamic instability;
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months prior to screening;
* Acute infection requiring intravenous antibiotics at the time of screening;
* Uncontrolled bleeding and coagulation disorders;
* Uncontrolled diabetes mellitus: IDDM or NIDDM;
* HIV positive or any other immunosuppressive disorder;
* Subject objects to the study protocol;
* Concurrent participation in any other clinical study;
* Physician objection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: asthmatic subjects or healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Study success will be declared if one of the following is met: A correlation of at least 0.25 (R2=0.25) will be found between WR and FEV1 measurements; A correlation of at least 0.7 will be found between clinical parameter and WZ measurements. | 6 months

SECONDARY OUTCOMES:
Evaluation of the safety of using the PulmoTrack® 2010 with WIM-PC™ Technologies for wheeze detection. Safety will be established by lack of adverse events. Since this is a Non Significant Risk (NSR) device serious adverse events are not expected | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Noam Gavriely, Prof., Study Director
Locations (1):
- Bnei-Zion Medical Center, Haifa, Israel